CLINICAL TRIAL: NCT00426985
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group Phase III Study of the Efficacy, Tolerability and Safety of Ketoprofen Topical Patch, 20% (KTP) in the Treatment of Pain Associated With Tendonitis or Bursitis of the Shoulder, Elbow or Knee
Brief Title: Efficacy and Safety of Ketoprofen Topical Patch 20% in the Treatment of Pain Associated With Shoulder, Elbow or Knee Tendonitis or Bursitis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sufficient number of subjects accrued to conduct analysis
Sponsor: Endo Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EN3269-304
Record Dates: First submitted 2007-01-24; First posted 2007-01-26 (Estimated); Last update posted 2008-08-14 (Estimated); Status verified 2008-08

CONDITIONS: Tendonitis; Bursitis
Keywords: Tendonitis; Bursitis; Pain; Shoulder Pain; Elbow Pain; Knee Pain; Tendon Injury; Muscle, Bone and Cartilage Disorders
MeSH Terms: conditions — Tendinopathy; Bursitis; Pain; Shoulder Pain; Tendon Injuries; Cartilage Diseases

INTERVENTIONS:
Drug: Ketoprofen Topical Patch 20%

SUMMARY:
The purpose of this study is to evaluate the effect of a ketoprofen topical patch on the pain associated with tendonitis or bursitis of the shoulder, elbow or knee

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled, parallel group study will be conducted in patients with tendonitis or bursitis of the shoulder, elbow or knee. Eligible patients will have tendonitis or bursitis or the shoulder, elbow or knee and will be randomized (1:1 ratio) to receive double-blind treatment with either the KTP or a matching placebo patch to be applied once daily for 21 days. Patients will return to the clinic for assessments on Day 3, Day 7, Day 14 and Day 21; a follow-up assessment will be conducted by telephone on Day 35. At each visit through Day 21, patients will rate their average pain intensity during daily activities and while at rest using the 11-point scale (range 0 to 10), and will rate their functional disability. Patients will also complete an electronic diary in which pain intensity and pain relief ratings will be recorded three times daily. The use of study treatment and rescue medication will be recorded in the diary each day. Ibuprofen will be provided as prn rescue medication.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 18 years of age or older
* Diagnosis of tendonitis or bursitis of the shoulder, elbow or knee
* Meet pain entry criteria
* Willing to discontinue use of any pain medication not provided by study

Exclusion Criteria:

* Have tendonitis or bursitis secondary to a systemic inflammatory disease, calcification or requiring surgery
* Have received corticosteroids in the 30 days preceding screening
* Have a history or physical examination finding that is incompatible with safe participation in the study
* Have a history or physical examination finding that is incompatible with study product use
* Are taking medications or other substances contraindicated due to the nature of the study medication or the potential for drug interactions.
* Are taking medications that may significantly affect renal function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2007-01; Primary Completion 2008-05 (Actual); Study Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
Average pain intensity during daily activities

SECONDARY OUTCOMES:
Average pain intensity while at rest; use of prn rescue medication; patient's and physician's global assessments of study medication, MPI, Sleep

CONTACTS AND LOCATIONS:
Overall Officials: PPD, Study Director — PPD Development, LP
Locations (1):
- PPD, Austin, Texas, United States